CLINICAL TRIAL: NCT03691259
Title: Examining the Effects of Ballet Training on Postural Stability in Older Adults
Brief Title: Effects of Ballet Training on Postural Stability in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1809-742
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Older Adults
Keywords: Dance; Postural stability; Ballet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance Group (Experimental): Dance group will participate in one-hour ballet classes twice per week for 10 weeks
  Interventions: Other: Ballet Classes
- Control Group (No Intervention): The control group will not participate in the ballet classes

INTERVENTIONS:
Other: Ballet Classes — Ballet classes will consist of learn the basic positions and combinations used in ballet, including: Plié, Tendu, Degagé, Rond de Jambe, Frappé, Chassé, Sauté, Pas de Bourrée, Glissade, and Révérance. Additional ballet movements and patterns may be employed as well.
  Arms: Dance Group

SUMMARY:
The purpose of this study is to examine the changes in postural stability in older adults following exposure to a beginning ballet dance technique course. Postural stability will be assessed at baseline and following the intervention using Wii Balance Boards as an affordable alternative to force plates. It is hypothesized that a significantly reduced body sway will be observed in participants following a ballet dance training course over a 10-week period.

DETAILED DESCRIPTION:
Postural stability (balance) is an essential skill across many genres of dance in order to create and maintain specific positions and motions with proper technique. Previously, it has been shown that dance interventions can lead to improvements in postural stability in elderly populations. However, there is limited research examining changes in balance following ballet dance class interventions for older adults.

One-hour ballet classes will be held twice per week in one of the two dance studios at Skidmore College. A dance student will serve as the lead teacher for each dance class session throughout the 10 weeks of ballet classes. Each week the participants will partake in 120 minutes of ballet dance training, starting with warm-up exercises at the barre and then working towards learning combinations in the center. They will learn the basic positions and combinations used in ballet, including: Plié, Tendu, Degagé, Rond de Jambe, Frappé, Chassé, Sauté, Pas de Bourrée, Glissade, and Révérance. Additional ballet movements and patterns may be employed as well. Skidmore students acting as teachers for the ballet classes will receive training packets with all necessary information about the logistics of the class and suggestions on how to be assist during the classes. The packet will discuss appropriate interactions and confidentiality during the class.

To assess postural stability, participants will be asked to stay in a static standing position for trials of 30 seconds while standing on a Wii board in four of the following conditions : 1) bilateral stance with eyes open, 2) bilateral stance with eyes closed, 3) unilateral stance on the right limb 4) unilateral stance on the left limb. Participants will be given a 15 seconds rest period between each trial and will be told they may stop and rest at any moment during the testing process. Data collection will take place at the multipurpose room (Williamson Sports Center), the intramural gym (Williamson Sports Center), or at the Prestwick Chase facility or the Saratoga Senior Center (if requested by an activities director) prior to the start of the ballet classes with post-testing to be completed the week of, or following, the final ballet class. Tests of postural stability will be verbally explained/instructed to create clear expectations for the test and to help decrease any fear or anxiety surrounding the process.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include being at least 55 years of age, independence with activities of daily living, and being free from cardiovascular or neurological disease

Exclusion Criteria:

* Exclusion criteria will include active participation in a physical therapy program with the goal of improving functional mobility, receiving dance training in the past, and requiring a walking aide
* For the experimental group only: missing six or more of the ballet classes offered during the 10-week period

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Postural Stability | 10 weeks
  Postural stability will be assessed through examination of average center of pressure velocity and maximum deviation from the mean

CONTACTS AND LOCATIONS:
Overall Officials: Sarah DiPasquale, DPT, Principal Investigator — Skidmore College
Locations (1):
- Skidmore College, Saratoga Springs, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT03691259/Prot_SAP_ICF_000.pdf